CLINICAL TRIAL: NCT05038449
Title: An IIT, Randomized, Single-Center, Open-Lable, Standard Therapy Controlled Study to Evaluate the Efficacy and Safety of Colchicine Tablets in Patients With COVID-19
Brief Title: Study to Evaluate the Efficacy and Safety of Colchicine Tablets in Patients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Public Health Clinical Center (Other Government)
Collaborators: Kunming Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Hongzhou Lu, Co-Director of Shanghai Public Health Clinical Center affiliated to Fudan University, Shanghai Public Health Clinical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KPC/QSXJ/01
Record Dates: First submitted 2021-09-05; First posted 2021-09-09 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Colchicine
Keywords: COVID-19; Colchicine Tablets; IIT Study
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine group (Experimental): The colchicine treatment includes an initial dose of 1 mg (1 mg and 0.5 mg two hours after), followed by 0.5 mg every 12 hours during the next 6 days and 0.5 mg every 24 hours until the completion of 10 days of total treatment.
  + standard therapy for COVID-19 according to the Novel Coronavirus Pneumonia Diagnosis and Treatment Plan (Trial 8th Edition).
  Interventions: Drug: Colchicine Tablets; Drug: Standard therapy
- Standard therapy group (Placebo Comparator): Standard therapy for COVID-19 according to the Novel Coronavirus Pneumonia Diagnosis and Treatment Plan (Trial 8th Edition).
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: Colchicine Tablets — Colchicine Tablets (Each tablet contains colchicine 0.5mg)
  Arms: Colchicine group
Drug: Standard therapy — Standard therapy for COVID-19 according to the Novel Coronavirus Pneumonia Diagnosis and Treatment Plan (Trial 8th Edition)

SUMMARY:
This study is designed for single-center, randomized, open label, standard therapy controlled. 60 COVID-19 subjects with a treatment period of 10 days and follow-up until 28 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of signing ICF, the subjects were 18 to 65 years old (including 18 and 65 years old), both men and women;
2. Within 72 hours before screening, any samples confirmed by the laboratory were positive for SARS-CoV-2;
3. Clinical classification was ordinary type according to the Novel Coronavirus Pneumonia Diagnosis and Treatment Plan (Trial 8th Edition)；
4. Symptoms appeared ≤ 5 days before randomization; Such as fever, cough, shortness of breath, sore throat and diarrhea;
5. Subjects were able to communicate well with the investigator, and understand and comply with the requirements of this study, understand and sign the ICF.

Exclusion Criteria:

1. Severe type patients who comply with any of the following：

   * Shortness of breath, RR ≥ 30 times/min;
   * In the resting state, the oxygen saturation is less than or equal to 93%;
   * Arterial oxygen partial pressure (PaO2)/oxygen inhalation concentration (FiO2) ≤ 300 mmHg (1mmHg=0.133kPa). Note: At high altitudes (above 1000 m), PaO2/FiO2 shall be corrected according to the following formula: PaO2/FiO2 × [760/atmospheric pressure (mmHg)];
   * Pulmonary imaging shows that patients with obvious lesion progression > 50% within 24-48 hours.
2. Critical type patients who comply with any of the following：

   * Respiratory failure occurs and mechanical ventilation is required;
   * Shock;
   * ICU monitoring and treatment are required for other organ failure.
3. People who are known to be allergic to the test drug and its components;
4. People with inflammatory bowel disease, chronic diarrhea, malabsorption;
5. People with previous neuromuscular disease;
6. People with severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2);
7. People with medical history of liver cirrhosis, active chronic hepatitis, or severe liver disease with serum GOT or GPT 3 times higher than the normal upper limit;
8. Patients who are taking colchicine or have a history of colchicine treatment (mainly chronic prescriptions for familial Mediterranean fever or gout);
9. People who have used immunosuppressants, corticosteroids, interleukin-1 inhibitors, or interleukin-6 inhibitors within 30 days before screening;
10. People who test positive for anti-SARS-CoV-2 immunoglobulin G (IgG);
11. People who have been vaccinated against COVID-19;
12. Any comorbidities that require surgery within 7 days before screening, or life-threatening comorbidities within 30 days before screening;
13. Suffering from malignant tumor diseases (excluding malignant tumors that have been cured and have not recurred in the past 5 years, completely resected basal cell and squamous cell skin cancers, and any type of cancer in situ that has been completely resected);
14. Suffering from any serious concomitant systemic disease, condition or disorder that the researcher believes should be prevented from participating in this study;
15. Pregnant or lactating women who have a positive human chorionic gonadotropin (hCG) test;
16. People who have a fertility plan or do not consent to effective non-drug contraception during the signing of the ICF to 6 months after the end of the trial;
17. Participated in other clinical studies within 30 days before screening;
18. People who have other factors that the researcher believes are not suitable for inclusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-06 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Recovery rate of clinical symptoms (fever, cough, expectoration, chest tightness, shortness of breath, dyspnea) and virus negative conversion rate (RT-PCR) at day 7 | Day 7

SECONDARY OUTCOMES:
Changes in the patients' clinical status through the WHO Clinical Progression Scale (scores 0-10) at day 7 | Day 7
  The scale provides a measure of illness severity across a range from 0 (not infected) to 10 (dead)
Changes in the patients' clinical status through the WHO Clinical Progression Scale (scores 0-10) at day 10 | Day 10
  The scale provides a measure of illness severity across a range from 0 (not infected) to 10 (dead)
Ventilator usage rate, usage time at day 7 | Day 7
Ventilator usage rate, usage time at day 10 | Day 10
Recovery rate and virus negative conversion rate (RT-PCR) of 10-day clinical symptoms (fever, cough, sputum expectoration, chest tightness, shortness of breath, dyspnea) | Day 10
Time for the virus negative conversion (RT-PCR) | Up to day 28
Time for observation in hospital | Up to day 28
Length of hospital stay | Up to day 28
Number of days in the intensive care unit | Up to day 28
Changes in inflammatory markers at day 7: C-reactive protein | Day 7
Changes in inflammatory markers at day 10: C-reactive protein | Day 10
Changes in inflammatory markers at day 7: TNF-alfa | Day 7
Changes in inflammatory markers at day 10: TNF-alfa | Day 10
Changes in inflammatory markers at day 7: IL-6 | Day 7
Changes in inflammatory markers at day 10: IL-6 | Day 10
Changes in inflammatory markers at day 7: IL-1β | Day 7
Changes in inflammatory markers at day 10: IL-1β | Day 10
Changes in severity markers at day 7: D-dimer | Day 7
Changes in severity markers at day 10: D-dimer | Day 10
Changes in myocardial damage at day 7: hs-cTn | Day 7
Changes in myocardial damage at day 10: hs-cTn | Day 10
Changes in myocardial damage at day 7: NT-proBNP | Day 7
Changes in myocardial damage at day 10: NT-proBNP | Day 10

CONTACTS AND LOCATIONS:
Overall Officials: Hongzhou Lu, PI, Principal Investigator — Shanghai Public Health Clinical Center
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No